CLINICAL TRIAL: NCT07362095
Title: An Exploratory Study on the Safety and Efficacy of Luspatercept in the Treatment of Anemia Following Allogeneic Hematopoietic Stem Cell Transplantation for Acute Leukemia
Brief Title: Luspatercept for the Treatment of Anemia Following Allogeneic Hematopoietic Stem Cell Transplantation(Allo-HSCT)
Acronym: Allo-HSCT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Liang Zhao, Professor, Zhujiang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-KY-242
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Acute Leukemia
Keywords: Acute leukemia; Allo-HSCT; Anemia; Luspatercept
MeSH Terms: conditions — Anemia | interventions — luspatercept

STUDY DESIGN:
Intervention Model Description: Luspatercept
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single-Arm Group (Experimental): All participants receive subcutaneous luspatercept at 1 mg/kg on day +7 and day +28 post-transplantation.
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — Study Treatment and Dosing Schedule According to the protocol, subcutaneous injections will be administered at a dose of 1 mg/kg on day +7 and day +28 post-transplantation. Inject into the upper arm, thigh, or abdomen. Doses requiring a larger volume (>1.2 mL) should be divided into similar volumes in separate syringes and injected at different sites. Use a new syringe and needle for each separate injection.
  Missed Dose: A dosing window of ±3 days is allowed, i.e., within day +7 ±3 days and day +28 ±3 days post-transplantation. If delayed, administer as soon as possible and continue with the regular dosing schedule (maintaining at least a 3-week interval between doses). If the ±3-day window is exceeded, the subject will be withdrawn from the study treatment.
  Other Names: Reblozyl®

SUMMARY:
This is a single-center, single-arm, prospective exploratory study designed to evaluate the safety and efficacy of luspatercept for the treatment of anemia following allogeneic hematopoietic stem cell transplantation in patients with acute leukemia. A total of 46 eligible subjects are planned to be enrolled. The primary efficacy endpoint is the proportion of patients achieving a hemoglobin increase of ≥1.5 g/dL at 8 weeks post-transplantation (without transfusion support) compared to baseline (the average of 3 days prior to the first dose). Secondary endpoints include assessing the impact of luspatercept on time to hematopoietic engraftment (neutrophil and platelet) and recording safety indicators such as adverse events, graft-versus-host disease, and infections. Subjects will receive subcutaneous luspatercept at 1 mg/kg on day +7 and day +28 post-transplantation.

DETAILED DESCRIPTION:
This is a single-center, single-arm, prospective, exploratory clinical study. The study plans to enroll 46 acute leukemia patients who have undergone allo-HSCT. All enrolled subjects will receive subcutaneous luspatercept at a dose of 1 mg/kg on day +7 (±3 days) and day +28 (±3 days) post-transplantation.

Study Procedures:

The study includes a screening period, treatment follow-up visits (for drug administration), and observation follow-up visits. Intensive follow-up within 2 months post-transplant includes assessments of vital signs, physical examinations, serial hematological and biochemical tests, transfusion records, engraftment status, T-lymphocyte subset analysis (day 28), and disease-related evaluations (e.g., minimal residual disease testing, week 8). Adverse events will be continuously monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed with acute leukemia.
2. Has undergone allogeneic hematopoietic stem cell transplantation (allo-HSCT).
3. Expected to survive for more than 3 months from the date of signing the informed consent form.
4. Willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures, and has provided written informed consent.
5. Women of childbearing potential must have a negative serum pregnancy test within prior to enrollment. Female subjects who are surgically sterile or postmenopausal for at least 2 years are considered not of childbearing potential. Male and female subjects of reproductive potential must agree to use effective contraception throughout the study period.
6. Hemoglobin (Hb) level < 80 g/L.

Exclusion Criteria:

1. Inadequate organ function, defined as:

1. Creatinine clearance < 60 mL/min;
2. Left ventricular ejection fraction (LVEF) < 55%;
3. Oxygen saturation (SpO₂) < 92% on room air;
4. Total bilirubin > 2 × the upper limit of normal (ULN);
5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 × ULN. 2. Poorly controlled hypertension, defined as repeated systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg despite adequate antihypertensive therapy, or a history of hypertensive crisis or hypertensive encephalopathy.

3. History of other malignancies (except for acute leukemia), unless the subject has been disease-free for ≥5 years. However, subjects with the following history/concomitant conditions are eligible:

1. Basal or squamous cell carcinoma of the skin;
2. Carcinoma in situ of the cervix;
3. Carcinoma in situ of the breast;
4. Incidental histological finding of prostate cancer (T1a or T1b as defined by the TNM staging system);
5. Solid tumors considered by the investigator to have no other known active disease.

4. Major surgery within 8 weeks prior to enrollment. The subject must have fully recovered from any prior surgery.

5. History of cerebrovascular accident (including ischemic, embolic, and hemorrhagic), transient ischemic attack, deep vein thrombosis (including proximal and distal), pulmonary or arterial embolism, arterial thrombosis, or other venous thrombosis within 6 months prior to enrollment. Note: Prior superficial thrombophlebitis is not an exclusion criterion.

6. Uncontrolled epilepsy, history of cerebral ischemia/hemorrhage, cerebellar disease, or other active central nervous system disorders.

7. Cardiac disease within 6 months prior to enrollment, including: myocardial infarction, uncontrolled angina, acute decompensated heart failure, New York Heart Association (NYHA) Class III-IV heart failure, or uncontrolled arrhythmia (as determined by the investigator).

8. Uncontrolled active systemic fungal, bacterial, or viral infection. 9. Evidence of human immunodeficiency virus (HIV) infection, active hepatitis B, and/or active hepatitis C.

10. History of pure red cell aplasia (PRCA) and/or anti-erythropoietin antibody.

11. Any condition or concomitant medication that may interfere with the interpretation of study data.

12. Known hypersensitivity to luspatercept or any of its excipients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with reduced transfusion requirement | 8 weeks post-Allo-HSCT (without transfusion support) compared to the pre-first-dose baseline (average Hb level from the three days prior to the first dose).
  Proportion of patients achieving an increase in Hb of ≥1.5 g/dL at 8 weeks post-Allo-HSCT (without transfusion support) compared to the pre-first-dose baseline (average Hb level from the three days prior to the first dose).

SECONDARY OUTCOMES:
Time to Granulocyte Engraftment | One month after allo-HSCT (i.e., 3 weeks after the first dose)
  Time interval from the day of stem cell infusion to the first day of three consecutive days with an absolute neutrophil count (ANC) greater than 0.5 G/L.
Time to Platelet Engraftment | One month after allo-HSCT (i.e., 3 weeks after the first dose)
  Time interval from the day of stem cell infusion to the first day of three consecutive days with an absolute platelet count ≥40 × 10⁹/L.
Incidence of drug-related adverse reactions | From baseline through 2 months post-administration of Luspatercept
  Record the occurrence of all adverse events, including the event type, severity, time of onset, relationship to the drug, and management actions taken. Analyze the incidence of adverse reactions (possibly) related to the drug, and the incidence of Grade ≥3 adverse reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Liang, Doctor, Principal Investigator — Zhujiang Hosptial of Southern Medical University
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the trial, data will be made public through the publication of academic papers. The original data can be requested via email.
Supporting Information: Study Protocol
Time Frame: Upon trial completion